# **Study Title:** A Phase 2/3 Study to Evaluate the Safety and Efficacy of Dociparstat Sodium for the Treatment of Severe COVID-19 in Adults at High Risk of Respiratory Failure

NCT Number: NCT04389840

**Document Date:** 06 November 2020

# Post-Cohort 1 or 2 Lock Analyses - Shells



Sponsor Name: Chimerix, Inc

Protocol Number and Title: CMX-DS-004

A Phase 2/3 Study to Evaluate the Safety and Efficacy of Dociparstat Sodium for Treatment of Severe COVID-19 in Adults at High Risk of

Respiratory Failure

Final Protocol Date: Protocol Amendment 3, dated 06 Nov 2020

Syneos Health Project Code: 7015085

Author(s): Roland Wolf, PhD, Lead Biostatistician

Version 2.0

Version Date: 12 March 2021

#### **Notice of Confidential and Proprietary Information**

The information contained in this document is confidential belonging to Chimerix, Inc. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Chimerix, Inc. However, this document may be disclosed to appropriate Institutional Review Board and Ethics Committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, Syneos Health should be notified promptly.

Chimerix, Inc: CMX-DS-004





| APPROVALS | and ACKNOWLEDGE | EMENT OF REVIEW |
|---|---|---|
| | Syneos Health | |
| | Roland Wolf | Electronically signed by: Roland Wolf<br>Reason: I am the author<br>Date: Mar 15, 2021 17:27 GMT+1 |
| Roland Wolf, PhD Principal Biostatistician | Signature | Date (DD-Mmm-YYYY) |
| Andrea Wirth | Andrea Wirth | Electronically signed by: Andrea Wirth<br>Reason: I am the approver<br>Date: Mar 15, 2021 17:35 GMT+1 |
| Senior Principal Biostatistician | Signature | Date (DD-Mmm-YYYY |
| | Blake Allman | Electronically signed by: Blake Allman<br>Reason: I am the approver<br>Date: Mar 16, 2021 08:51 GMT |
| Blake Allman Principal Stat Programmer | Signature | Date (DD-Mmm-YYYY) |
| | Chimerix | |
| | Thomas M. | Digitally signed by Thomas M. Brundage |
| Thomas M. Brundage | Brundage | Date: 2021.03.15 11:30:00 -04'00' |
| Executive Director, Biostatistics | Signature | Date (DD-Mmm-YYYY) |

Syneos Health #7015085

Chimerix, Inc: CMX-DS-004





# **Revision History**

| Version # | Date<br>(dd-mmm-yyyy) | Document Owner | Revision Summary |
|---|---|---|---|
| 1.0 | 17 Sep 2020 | Roland Wolf | Initial Release Version |
| 2.0 | 12 Mar 2021 | Roland Wolf | Updated for Protocol Amendment 3. Clarify analysis of subjects randomized but not treated. |



# **TABLE OF CONTENTS**

# **List of Tables**

| Table 1: Demographics and Baseline Characteristics – Safety Set | 11 |
|---|---|
| Table 2: Listing of demographics, baseline characteristics, study drug usage and disposition – Safety Set | |
| Table 3: Study drug usage – Safety Set | 14 |
| Table 4: Listing of study drug interruptions / discontinuations – Safety Set 1 | 15 |
| Table 5: Treatment disposition – Safety Set | 16 |
| Table 6: Study disposition – Randomized Subjects | 17 |
| Table 7: Proportion of subjects who go on invasive mechanical ventilation or ECMO - Safety Set | 18 |
| Table 8: Treatment-emergent Adverse Events (TEAEs) – Safety Set | 21 |
| Table 9: Severe, life-threatening or fatal treatment emergent Adverse Events – Safety Set | 22 |
| Table 10: Treatment emergent Adverse Events leading to study drug discontinuation – Safety Set | 22 |
| Table 11: Serious treatment emergent Adverse Events – Safety Set | 22 |
| Table 12: Listing of Serious Adverse Events and Adverse Events of Special Interest – Safety Set | 23 |
| Table 13: Overview CTCAE v5.0 Grades | 24 |
| Table 14: Distribution of laboratory grade by parameter and visit – Safety Set 2 | 25 |
| Table 15: Listing of laboratory results – Safety Set | 26 |
| Table 16: Shift-table of laboratory results – Safety Set | 27 |
| Table 17: Listing of Prior and Concomitant Medications (only Targeted Medications) – Safety Set | 30 |
| Table 18: Proportion of and time to invasive mechanical ventilation or all-cause mortality – ITT Set | 33 |
| Table 19: Proportion of and time to all-cause mortality – ITT Set | 35 |
| Table 20: Proportion of participants who are alive, discharged from the hospital, and not using home oxygen – ITT Set | |

# Syneos Health #7015085

Chimerix, Inc: CMX-DS-004



Post-Cohort 1 or 2 Lock Analysis Shells: Version 2.0, dated 12 March 2021

| Table 21: Clinical status assessed by the NIAID ordinal scale at fixed tin | - |
|---|---|
| Table 22: Time to clinical improvement – ITT Set | 40 |
| Table 23: Number of ventilator-free days from baseline through Day 28 | |
| Table 24: Time to last hospital discharge – ITT Set | 43 |
| Table 25: Time to first hospital discharge – ITT Set | 45 |
| List of Figures | |
| Figure 1: Time to first invasive mechanical ventilation or ECMO (KM-I Safety Set | |
| Figure 2: Duration of first invasive mechanical ventilation or ECMO (K Safety Set | |
| Figure 3: Selected laboratory parameters over time (Box-Whisker-Plot) Set | |
| Figure 4: Biomarkers during the course of the study – Safety Set | 31 |
| Figure 5: Time to invasive mechanical ventilation, ECMO or all-cause r (KM-Plot) – ITT Set | |
| Figure 6: Time to all-cause mortality (KM-Plot) – ITT Set | 36 |
| Figure 7: Time to clinical improvement (KM-Plot) – ITT Set | 41 |
| Figure 8: Time to last hospital discharge (KM-Plot) – ITT Set | 44 |
| Figure 9: Time to first hospital discharge (KM-Plot) – ITT Set | 45 |

Syneos Health #7015085

Chimerix, Inc: CMX-DS-004





# 1. PURPOSE

This is a randomized, double-blind, placebo-controlled, Phase 2/3 study to determine the safety and efficacy of dociparstat in adults with acute lung injury associated with severe COVID-19 who are at high risk of respiratory failure.

An independent unblinded data monitoring committee (DMC) will review safety data from Cohort 1 to make a recommendation on dose escalation in Cohort 2 and review safety data from both Cohorts 1 and 2 to make a recommendation on dosing in Cohort 3. The sponsor will consider the DMC recommendation when determining the actual doses for Cohorts 2 and 3.

Due to the evolving standard of care for COVID-19, the sponsor may decide to unblind and review study data following Cohorts 1 and/or 2.

The purpose of this document is to describe the pre-defined post-Cohort 1 or 2 lock analysis. This document specifies the derivations and TFL package and is based on the study protocol amendment 3, dated 06 November 2020.

Chimerix, Inc: CMX-DS-004





# 2. INTRODUCTION

Cohort 1 contains 6 participants randomized to dociparstat, 6 randomized to placebo. Dociparstat will be dosed as 4 mg/kg IV bolus followed by continuous infusion of 0.25 mg/kg/hr.

Cohort 2 includes 6 participants randomized to dociparstat, 6 randomized to placebo. Dociparstat will be dosed as 4 mg/kg IV bolus followed by continuous infusion of 0.325 mg/kg/hr (dose to be confirmed after review of data from Cohort 1).

Based on Protocol Amendment 3, dated 06 November 2020, the randomization ratio (dociparstat: placebo) changed from 1:1 in Cohort 1 to 2:1 in the following cohorts.

Both Cohorts 1 and 2 may be unblinded to the entire team following cleaning and database lock of Cohort 1/2 data. The full randomization code will remain blinded as is; in this event, only the Cohort 1/2 assignments will be unblinded.

The first part of the analysis defined in this document will be eqivalent to the statistical output delivered to the DMC-members for the 2nd Cohort (see Section 5.1), however with all data collected until End of Study (EOS).

Post-Cohort 1 or 2 Lock Analysis Shells: Version 2.0, dated 12 March 2021



# 3. DERIVATIONS AND DEFINITIONS

#### Kaplan-Meier estimates

Time to xxx (days): Days are calculated as (start date/time – first study drug date/time)/24h). Time will be censored at last individual date/time reported.

Worst-case results in 2 scenarios for missing time-values:

1. Missing time for negative events will be imputed with "00:01", missing time for censored observations will be imputed with "23:59".

Negative events are:

- Time to first invasive mechanical ventilation or ECMO
- Time to first invasive mechanical ventilation, ECMO or all-cause mortality
- Time to all-cause mortality
- 2. Missing time for positive events will be imputed with "23:59", missing time for censored observations will be imputed with "00:01".

Positive events are:

- Time to clinical improvement
- Time to hospital discharge

In addition, to avoid bias in the positive events, deaths occurring prior to the positive event being observed will censored at Day 28.

#### Ventilator-free days

Ventilator-free days are only counted from baseline through Day 28 or end of study, whichever comes first. They are derived based on the eCRF data collected on the Ventilator/Oxygen/Medical Care Status CRF page, Ventilator-free days are all days where Ventilator/Oxygen/Medical Care Status is not equal "Invasive Mechanical Ventilation or extracorporeal membrane oxygenation (ECMO)".

Ventilator days are defined as cumulative rounded number of days with Ventilator/Oxygen/Medical Care Status = "Invasive Mechanical Ventilation or extracorporeal membrane oxygenation (ECMO)" devided by 24 h. Missing time for start will be imputed with "00:01", missing time for stop will be imputed with "23:59".

**Study duration in days is defined as**: Date of study completion (or date of early study discontinuation) – date of first study treatment + 1. For subjects randomized but not treated the date of randomization will be used instead of first study treatment date. The maximum study duration is set to 28 days, even if study completion or study discontinuation is after 28 days.

**Ventilator-free days are defined as**: study duration - number of ventilator days. For subjects who died during the course of the study, the number of ventilator-free days will be defined as 0.

Post-Cohort 1 or 2 Lock Analysis Shells: Version 2.0, dated 12 March 2021



# Randomized, but not treated subjects:

The following rules will apply for randomized subjects without receiving study treatment, if not stated otherwise:

- Calculations referring to start of treatment or baseline will be performed with respect to randomization date/time.
- Study duration in days is calculated as study discontinuation date randomization date +1.
- In Kaplan-Meier analysis the "time-to" will be censored at 0.

Chimerix, Inc: CMX-DS-004





#### 4. CONVENTIONS FOR SUMMARY TABLES AND LISTINGS

At the top of each table/listing/figure, the first three title lines should read:

```
Chimerix
CMX-DS-004
Post-Cohort 1/2 Lock Analysis - FINAL (Unblinded)
```

Following those titles, the next title should include the output number and a description of the table/listing content, including the Analysis Set used.

The next line is an optional sub-title with description of a subgroup, if applicable.

Horizontal lines will appear before and after the column heading of the table/listing. Footnotes will be put under the main body of text and each new footnote should start with a new line. Very long footnotes will be presented only on the very first page of the output.

At the bottom of each TFL, the following information should be printed: date of the data base cut off, date and time of the run of the TFL and name of the program.

```
Data Cut-off date: DDMMMYYYY;
Program name: M:\project-sas\chimerix\7015085\biostat\3-cohort\tables\production\xxxxx.sas
Run date: DDMMMYYYY HH:MM

Page X of Y
```

Outputs will be prepared in landscape layout unless otherwise specified. Blank margins of all tables and listings will be a minimum of 1 inch. In general, Courier New 8 point font will be used.

#### **Listings Layout**

Listings will contain the data of all subjects except when otherwise specified. The following visit labels will be used (shorthand in parentheses), but data will be sorted by assessment date (including the Unscheduled Visits):

- Screening (SCRN)
- o Baseline (D1)
- o Day 2 (D2)
- o Day 3 (D3)
- o Day 4 (D4)
- Day 5 (D5)
- Day 6 (D6)
- Day 7 (D7)
- o Day 8 (D8)
- o Day 14 (D14)
- o Day 28 (D28)
- o Early Tx DC (TXDC)
- Unscheduled (UNSCH)

# 5. TABLE SHELLS

# 5.1. DMC - TABLE SHELLS

Table 1: Demographics and Baseline Characteristics - Safety Set

| | DSTAT 0.25 | Cohort 1 PBO | DSTAT 0.325 | Cohort 2 PBO | Total |
|---|---|---|---|---|---|
| | N=xxx | N=xxx | N=xxx | N=xxx | N=xxx |
| Gender, n(%) | | | | | |
| Male | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Female | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Unknown/Not Answered | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Race, n(%) | | | | | |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/Not Answered | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n(%) | | | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/Not Answered | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Age (years) | | | | | |
| n | Xxx | xxx | xxx | xxx | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | Xx | xx | xx | xx | XX |
| Q1, Q3 | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | xx, xx |
| Age (years), n(%) | | | | | |
| < 60 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >=60 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Weight (kg) | | | | | |
| N | XXX | XXX | XXX | xxx | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | xx.x | xx.x | XX.X |
| Median | XX | XX | XX | XX | XX |
| Q1, Q3 | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |
| Min, Max | xx, xx | XX, XX | xx, xx | xx, xx | XX, XX |

Syneos Health #7015085, Chimerix, Inc, Protocol # CMX-DS-004, Post-Cohort 1 or 2 Lock Analysis Shells: Version 2.0, dated 12 Mar 2021

| | DSTAT 0.25 | Cohort 1 PBO | DSTAT 0.325 | Cohort 2 PBO | Total |
|---|---|---|---|---|---|
| | N=xxx | N=xxx | N=xxx | N=xxx | N=xxx |
| Height (cm) | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX | xx | xx | xx | XX |
| Q1, Q3 | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| Body mass index (kg/m2) | | | | | |
| n | xxx | xxx | XXX | xxx | XXX |
| Mean | xx.x | xx.x | XX.X | xx.x | XX.X |
| SD | xx.x | XX.X | XX.X | XX.X | XX.X |
| Median | XX | xx | xx | xx | XX |
| Q1, Q3 | xx, xx | xx, xx | xx, xx | xx, xx | XX, XX |
| Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX |
| Temperature (°C) | | | | | |
| n | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX | XX | XX | XX | XX |
| Q1, Q3 | XX, XX | xx, xx | xx, xx | xx, xx | XX, XX |
| Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Fever, n(%) | | | | | |
| <= 37.2°C | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| > 37.2°C to 38.2°C | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| > 38.2°C | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NIAID-Score (IRT), n(%) | | | | | |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NIAID-Score (actual), n(%) | | | | | |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; SD: Standard deviation; Q1, Q3: First, third quartile; Min: minimum; Max: maximum.

Page X of Y

Baseline is defined as last measurement prior to or on the date of first study treatment.

NIAID-Score (IRT): directly entered in RAVE by the investigator.

NIAID-Score (actual): calculated using hospitalization and ventilation status at time of randomization.

Table 2: Listing of demographics, baseline characteristics, study drug usage and disposition - Safety Set

| Subject<br>Age/Sex | Treatment<br>Group | Race | Ethni-<br>city | Weight<br>(kg) | BMI<br>(kg/m2) | Temp<br>(°C) | NIAID (IRT / actual) | Bolus received / # infusion days | Treatment disposition | Study<br>disposition | Death /<br>Date |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 999-999<br>/70/F | | Asian | HL | xx.x | | XX.X | 4 / 4 | Yes / 3 | Discontinued:<br>AE | Discontinued:<br>Progression | |
| 999-999<br>xx/xx | Cohort 1 PBO | Other: xxxxxx | NHL | XX.X | XX.X | | 3 / 3 | Yes / 7 | Discontinued:<br>Other: xxx | Discontinued:<br>FUP | |
| 999-999<br>xx/xx | Cohort 1 PBO | Other: | NHL | xx.x | XX.X | | 3 / 3 | Yes / 7 | Completed | Completed | Yes /<br>ddMMMYYY |
| 999-999<br>xx/xx | Cohort 1 PBO | Other: xxxxxx | NHL | XX.X | XX.X | | 3 / 4 | Yes / 7 | Unknown | Ongoing | |

Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino

NIAID-Score (IRT): directly entered in RAVE by the investigator.

NIAID-Score (actual): calculated using hospitalization and ventilation status at time of randomization.

Page X of Y

#### (Notes for programmer:

- Sorted by subject number
- -Disposition: Progression=Progression of disease, AE=Adverse Event, Prohibited=Patient requires use of a prohibited therapy, Compliance=Non-compliance, FUP=Lost to follow-up, Consent=Patient withdrawal of consent, Physician=Physician decision, Sponsor=Sponsor decision, Improvement=Improvement of condition under study, UNK=Unknown/Not answered)

Table 3: Study drug usage - Safety Set

| | DSTAT 0.25<br>N=xxx | Cohort 1 PBO<br>N=xxx | DSTAT 0.325<br>N=xxx | Cohort 2 PBO<br>N=xxx |
|---|---|---|---|---|
| Bolus received, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Infusion (days received), n(%) | | | | |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; Infusion (days received): Study drug administered at any time during the corresponding study-day (cumulated).

Page X of Y

Table 4: Listing of study drug interruptions / discontinuations - Safety Set

| Subject<br>Age/Sex/Race | Treatment<br>Group | Visit | Start<br>Date / Time | Stop<br>Date / Time | Bolus /<br>Infusion no | Total Voulume<br>Given (mL) | Interrupted due to | Permanently discontinued due to |
|---|---|---|---|---|---|---|---|---|
| 999-999 /<br>69/F/W | DSTAT 0.25 | Baseline (D1) | ddMMMyy hh:mm | ddMMMyy hh:mm | Bolus | 999.99 | Adverse Event | |
| | | Day 2 (D2)<br>Day 3 (D3)<br>Day 4 (D4) | ddMMMyy hh:mm<br>ddMMMyy hh:mm<br>ddMMMyy hh:mm<br>ddMMMyy hh:mm | ddMMMyy hh:mm<br>ddMMMyy hh:mm<br>ddMMMyy hh:mm<br>ddMMMyy hh:mm | 1<br>2<br>3<br>4 | 999.99<br>999.99<br>999.99<br>999.99 | Other:xxxxxx | Adverse Event<br>Other: xxxxxx |
| 999-999 /<br>35/M/B | Cohort 1 PBO | Baseline (D1) | ddMMMyy hh:mm | ddMMMyy hh:mm | Bolus | 999.99 | Adverse Event | |
| | | Day 2 (D2) | ddMMMyy hh:mm<br>ddMMMyy hh:mm | ddMMMyy hh:mm<br>ddMMMyy hh:mm | 1<br>2 | 999.99<br>999.99 | | |

Page X of Y

(Note for programmer: Sorted by subject number, start date, start time)

Table 5: Treatment disposition - Safety Set

| Treatment disposition | | | | |
|---|---|---|---|---|
| Primary reason for treatment discontinuation | DSTAT 0.25 | Cohort 1 PBO | DSTAT 0.325 | Cohort 2 PBO |
| | N=xxx | N=xxx | N=xxx | N=xxx |
| Commisted to the commist of (0) | ( | /> | / | () |
| Completed treatment, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Treatment disposition unknown, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued treatment, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for treatment discontinuation, n(%) | | | | |
| Progression of disease | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient requires use of a prohibited therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-compliance | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patient withdrawal of consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Physician decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sponsor decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Improvement of condition under study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/Not Answered | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death (during treatment period) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N;

Page X of Y

(Note for programmer: Death (during treatment period) to be derived in case death date = date of last treatment start date or stop date)

Table 6: Study disposition - Randomized Subjects

| Study Disposition | | | | |
|---|---|---|---|---|
| Primary reason for early termination | DSTAT 0.25 | Cohort 1 PBO | DSTAT 0.325 | Cohort 2 PBO |
| | N=xxx | N=xxx | N=xxx | N=xxx |
| Randomized subjects, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Randomized not treated subjects, n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Treated subjects, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Completed study, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ongoing, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued study | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary reason for study discontinuation, n(%) | | | | |
| Patient withdrawal of consent | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Adverse Event | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Use of a prohibited therapy | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Non-compliance | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sponsor decision | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown/Not Answered | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death, n(%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of randomized subjects in a specific group; n = Number of subjects with data available; Percentages are based on N;

Page X of Y

Table 7: Proportion of subjects who go on invasive mechanical ventilation or ECMO - Safety Set

| | DSTAT 0.25 | Cohort 1 PBO | DSTAT 0.325 | Cohort 2 PBO |
|---|---|---|---|---|
| | N=XXX | N=xxx | N=xxx | N=xxx |
| Number of subjects with any invasive | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| mechanical ventilation, ECMO or early study discontinuation, n (%) (a) | | | | |
| Any invasive mechanical ventilation | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Early study discontinuation < Day 25 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Kaplan-Meier estimates (b) | | | | |
| Number of censored subjects, n (%) (b) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to first invasive mechanical | | | | |
| ventilation or ECMO (days) (b) | | | | |
| 25% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| Median (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| 75% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| Number of subjects who stopped invasive mechanical ventilation or ECMO, $n(%)$ (c) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Kaplan-Meier estimates (c) | | | | |
| Number of censored subjects, n (%) (c) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Duration of first invasive mechanical | | | | |
| ventilation or ECMO (days) (c) | | | | |
| 25% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| Median (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| 75% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; ECMO: Extracorporeal membrane oxygenation.

<sup>(</sup>a) Subjects with any invasive mechanical ventilation, ECMO or early study discontinuation before Day 25 will be counted as event.

<sup>(</sup>b) Kaplan-Meier estimates: Subjects with any invasive mechanical ventilation or ECMO will be counted as event. All other subjects will be censored. Time to first invasive mechanical ventilation or ECMO (days): Days are calculated as (start date/time - first study drug date/time)/24h). Time will be censored at last individual date/time reported. If time is not available for events "00:01" will be imputed, for censored observations "23:59" will be imputed.

<sup>(</sup>c) Kaplan Meier estimates: Duration of first invasive mechanical ventilation or ECMO (days): Only calculated for subjects with an invasive mechanical ventilation or ECMO reported. Duration is calculated as (stop date/time - start date/time)/24h). If start time is not available "00:01" will be imputed, if end time is missing "23:59" will be imputed. Duration will be censored for subjects with ongoing ventilation at last individual date/time reported.

Page X of Y

Figure 1: Time to first invasive mechanical ventilation or ECMO (KM-Plot) - Safety Set

Kaplan-Meier Plot: y-axis: range: 0% to 100% by 20% label: Event-free Probability reference-line: 50% x-axis: range: 0 to xxx (depending on data), by 7 days label: Time to Event (Days) Lines: solid different colors/line styles for the treatment-groups starting at (100%/Baseline) Censored values marked Please use the following footnote for Figure 1: N = Number of subjects in a specific group; (+) = censored values; Kaplan-Meier estimates: Subjects with any invasive mechanical ventilation or ECMO will be counted as event. All other subjects will be censored. Time to first invasive mechanical ventilation or ECMO (days): Days are calculated as (start date/time - first study drug date/time)/24h). Time will be censored at last individual date/time reported. If time is not available for events "00:01" will be imputed, for censored observations "23:59" will be imputed.

Figure 2: Duration of first invasive mechanical ventilation or ECMO (KM-Plot) - Safety Set

```
Kaplan-Meier Plot:
y-axis:
       range: 0% to 100% by 20%
       label: Event Probability
       reference-line: 50%
x-axis:
       range: 0 to xxx (depending on data), by 7 days
       label: Duration (Days)
Lines:
       solid
       different colors/line styles for the treatment-groups
       starting at (0%/Baseline)
       Censored values marked
Please use the following footnote for Figure 2:
N = Number of subjects in a specific group; (+) = censored values;
Kaplan Meier estimates: Duration of first invasive mechanical ventilation or ECMO (days): Only calculated for subjets with an
invasive mechanical ventilation of ECMO reported. Duration is calculated as (stop date/time - start date/time)/24h. If start time
is not available "00:01" will be imputed, if end time is missing, "23:59" will be imputed. Duration will be censored for subjects
with ongoing ventilation at last individual date/time reported.
```

Table 8: Treatment-emergent Adverse Events (TEAEs) - Safety Set

| Primary system organ class<br>Preferred term | DSTAT 0.25<br>N=xxx<br>n (%) | Cohort 1 PBO<br>N=xxx<br>n (%) | DSTAT 0.325<br>N=xxx<br>n (%) | Cohort 2 PBO<br>N=xxx<br>n (%) |
|---|---|---|---|---|
| Number (%) of subjects with at least one such AE | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| SOC 1 | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| PT 1 | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| PT 2 | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| : | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| SOC 2 | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| : | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |

N = Number of subjects in a specific group; n = Number of subjects with at least one event in the category; Percentages are based on N; Adverse events are coded using MedDRA version 23.0.

If a subject has multiple occurrences of an AE, the subject is presented only once in the respective subject count (n).

Page X of Y

(Note for programmer: AEs are sorted by decending patients' frequency of SOC and by decending frequency of PT within the SOC in the DSTAT 0.25)

Table 9: Severe, life-threatening or fatal treatment emergent Adverse Events - Safety Set

For the layout refer to Table 8

(Notes for programmer:
- Change first line in the table to "Number (%) of subjects with at least one such AE".
- TEAEs with the following AE severity grades are reported: Grade 3 (Severe), Grade 4 (Life-threatening), Grade 5 (Fatal).)

Table 10: Treatment emergent Adverse Events leading to study drug discontinuation - Safety Set

For the layout refer to Table 8

(Note for programmer: Change first line in the table to "Number (%) of subjects with at least one such AE".

For the layout refer to Table 8

(Note for programmer: Change first line in the table to "Number (%) of subjects with at least one such TEAE".

Table 12: Listing of Serious Adverse Events and Adverse Events of Special Interest - Safety Set

| Subject<br>Age/Sex/Race | Treatment<br>Group | Preferred term<br>Verbatim | Start Date<br>(Study Day) | Stop Date<br>(Study Day) | Severity | Relation-<br>ship | Outcome | Serious<br>AE | AE of Special<br>Interest | Action taken<br>with study drug |
|---|---|---|---|---|---|---|---|---|---|---|
| 999-999 /<br>70/F/W | DSTAT<br>0.25 | PT1<br>xxxxxxxxx | DdMMMyy (xx) | DdMMMyy (xx) | Mild | Related | Fatal | Yes | Yes | Discontinued |
| 999-999 /<br>xx/xx/xx | Cohort 1<br>PBO | PT1<br>xxxxxxxxx | DdMMMyy (xx) | DdMMMyy (xx) | Mild | Related | Recovered | No | Yes | No Change |

Note: Adverse events are coded using MedDRA version 23.0.

Study Days prior to first treatment date are calculated as (actual date - first treatment date), after first treatment date as (actual date - first treatment date) + 1.

Page 1 of x

(Notes for programmer:

- Sorted by subject number, start date, stop date, Preferred term and Verbatim
- Outcome: Ongoing=Not recovered (Ongoing), Sequelae=Recovered with Sequelae, Unknown=Unknown/Lost to Follow-up
- Action taken with study drug: Interrupted=Study drug temporarily interrupted, Discontinued=Study drug permanently discontinued)

Table 13: Overview CTCAE v5.0 Grades

| Parameter | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hemoglobin | <lln -="" 10.0="" dl<br="" g=""><lln -="" 6.2="" l<br="" mmol=""><lln -="" 100="" g="" l<="" td=""><td>&lt;10.0 - 8.0 g/dL<br/>&lt;6.2 - 4.9 mmol/L<br/>&lt;100 - 80g/L</td><td>&lt;8.0 g/dL<br/>&lt;4.9 mmol/L<br/>&lt;80 g/L</td><td>NA</td></lln></lln></lln> | <10.0 - 8.0 g/dL<br><6.2 - 4.9 mmol/L<br><100 - 80g/L | <8.0 g/dL<br><4.9 mmol/L<br><80 g/L | NA |
| Platelets | <lln -="" 75,000="" mm3;<br=""><lln -="" 10e9="" 75.0="" l<="" td="" x=""><td>&lt;75,000 - 50,000/mm3;<br/>&lt;75.0 - 50.0 x 10e9/L</td><td>&lt;50,000 - 25,000/mm3;<br/>&lt;50.0 - 25.0 x 10e9/L</td><td></td></lln></lln> | <75,000 - 50,000/mm3;<br><75.0 - 50.0 x 10e9/L | <50,000 - 25,000/mm3;<br><50.0 - 25.0 x 10e9/L | |
| Activated Partial Thromboplasting Time (aPTT) | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN | NA |
| Prothrombin Intl. Normalized Ratio (INR) | >1.2 - 1.5 | >1.5 - 2.5 | >2.5 | NA |
| Aspartate Aminotransferase (AST) | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Alanine Aminotransferase (ALT) | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN |
| Total Bilirubin | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN |
| Creatinine | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 6.0 x ULN | >6.0 x ULN |
| Creatinine Clearance, Estimated | <lln -="" 60="" min<="" ml="" td=""><td>&lt;60 - 30 ml/min</td><td>&lt;30 - 15 ml/min</td><td>&lt;15 ml/min</td></lln> | <60 - 30 ml/min | <30 - 15 ml/min | <15 ml/min |

Table 14: Distribution of laboratory grade by parameter and visit - Safety Set

Parameter: <Hemoglobin> <Platelets> <Activated partial thromboplastin time (aPTT)> <Prothrombin International Normalized Ratio (INR)> <Aspartate aminotransferase (AST)> <Alanine aminotransferase (ALT)> <Total bilirubin> <Creatinine> <Creatinine Clearance, Estimated >

| Scheduled Visit Grades (a) | DSTAT 0.25<br>N=xxx | Cohort 1 PBO<br>N=xxx | DSTAT 0.325<br>N=xxx | Cohort 2 PBO<br>N=xxx |
|---|---|---|---|---|
| Grades (a) | IV-AAA | IN-AAA | IN-AAA | IN-XXX |
| Baseline | | | | |
| Grade 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Maximum Post-baseline Grad | de | | | |
| Grade 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Grade 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Unknown | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; (a) CTCAE v5.0 grades using absolute thresholds without accounting for baseline.

Baseline value is defined as the last non-missing measurement prior to, or on the date/time of the first administration of study treatment.

NA = not applicable

Page X of Y

#### (Notes for programmer:

- CTCAE Grades: Unknown: missing result (or missing upper limit of normal for parameters requiring ULN for grading). Grade 0: any result not graded 1, 2, 3, 4 or Unknown.
- display only for visit Baseline and Maxiumum Grade per subject and all 6 categories (Grade 0 Grade 4 and Unknown), if applicable.
- generate a post-baseline Maximum Grade per subject (incl. unscheduled measurements)
- for the generation of Maxiumum Grade use the following order: Unknown Grade 0 Grade 1,.... Grade 4)
- Calculation of creatinine clearance (CC) (Cockcroft-Gault):

```
(140 - age \ (years)) 
 CC (ml/min) = ----- * baseline weight \ (kg) * (0.85 if female) 
 0.8143 * serum \ creatinine \ (\mu mol/L)
```

Table 15: Listing of laboratory results - Safety Set

| Subject<br>Age/Sex/Race | Treatment<br>Group | Parameter | Date/Time | Visit | Value \$ | | Unit | Lower<br>Limit | Upper<br>Limit | Grade<br>(a) |
|---|---|---|---|---|---|---|---|---|---|---|
| 999-999 | DSTAT 0.25 | Hemoglobin | Ddmmmyy/mm:hh | Screening | 99999 н | NCS | Unit | LLL | UUU | 1 |
| 70/F/W | | | Ddmmmyy/mm:hh | Baseline | 99999 L | CS | Unit | LLL | UUU | 4 |

(a) CTCAE v5.0 grades using absolute thresholds without accounting for baseline. Grade=0 and Grade=Unknown are not displayed. \$: H = Above upper limit of normal; L = Below lower limit of normal, NCS = Not clinically significant, CS= Clinically significant. Visit "Early Tx DC (TXDC)" denotes Early Treatment Discontinuation Visit.

#### (Notes for programmer:

- Sorted by subject number, Parameter, date and time
- The following parameter will be displayed: Hemoglobin, platelets, activated partial thromboplastin time (aPTT), prothrombin time (PT), prothrombin international normal ratio (INR), d-dimer, Anti-Xa, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, creatinine, Creatinine Clearance, Estimated.
- LLN for creatinine clearance is fixed 90 mL/min
- CTCAE Grades: reference Table 13.)

Table 16: Shift-table of laboratory results - Safety Set

Parameter: <Hemoglobin> <Platelets> <Activated partial thromboplastin time (aPTT)> <prothrombin time (PT)> <Prothrombin International Normalized Ratio (INR)> <d-dimer> <Anti-Xa> <Aspartate aminotransferase (AST)> <Alanine aminotransferase (ALT)> <Total bilirubin> <Creatinine> <Creatinine Clearance, Estimated>

| | DSTAT 0.25<br>N=xxx | | | Baseline<br>Cohort 1 PBO<br>N=xxx | | | | (D1) DSTAT 0.325 N=xxx | | | Cohort 2 PBO<br>N=xxx | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | <lln< th=""><th>Normal</th><th>&gt;ULN</th><th></th><th>Normal</th><th>&gt;ULN</th><th><lln< th=""><th>Normal</th><th>&gt;ULN</th><th></th><th>Normal</th><th>&gt;ULN</th></lln<></th></lln<> | Normal | >ULN | | Normal | >ULN | <lln< th=""><th>Normal</th><th>&gt;ULN</th><th></th><th>Normal</th><th>&gt;ULN</th></lln<> | Normal | >ULN | | Normal | >ULN |
| Post-Baseline | | | | | | | | | | | | |
| Minimum, n(%) | | | | | | | | | | | | |
| <lln< td=""><td>XX</td><td>XX</td><td>xx</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td><td>XX</td></lln<> | XX | XX | xx | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Normal | XX | XX | xx | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| >ULN | XX | XX | xx | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Post-Baseline | | | | | | | | | | | | |
| Maximum, n(%) | | | | | | | | | | | | |
| <lln< td=""><td>XX</td><td>xx</td><td>xx</td><td>XX</td><td>XX</td><td>xx</td><td>XX</td><td>XX</td><td>xx</td><td>XX</td><td>XX</td><td>XX</td></lln<> | XX | xx | xx | XX | XX | xx | XX | XX | xx | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| Normal | XX | xx | xx | XX | XX | XX | XX | XX | xx | XX | XX | XX |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |
| >ULN | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx | xx |
| | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) | (xx.x) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; Normal: Within normal range, LLN: Lower limit of normal, ULN: Upper limit of normal.

Only subjects with baseline and at least one post-baseline value are considered.

Baseline value is defined as the last non-missing measurement prior to, or on the date/time of the first administration of study treatment. NA = not applicable.

Page X of Y

#### (Notes for programmer:

- generate a post-baseline Maximum Value and post-baseline Minimum Value per subject (incl. unscheduled measurements
- LLN for creatinine clearance is fixed 90 mL/min
- if ULN (eg CC) available, please display n/a

- )

Figure 3: Selected laboratory parameters over time (Box-Whisker-Plot) - Safety Set

Box-Whisker-Plots: by <Parameter> (<unit>), Cohort X, Reference Ranges xxx - yyyy <unit>
y-axis:
range: depending on data
label: Value

x-axis:
range: Visits: Screening, D1 to D28 (depending on data) visit. Incl Early Tx DC at the end of the x-axis.
label: Visit
Box-Whisker Plots:
different styles/colors for the treatment-groups

Plots shifted to not overlap
Default SAS Box-Whisker-Plots - Min, 25%, Median, 75%, Max. Whiskers as 1.5 IQR. Mean included.

Footnotes to be used for the Box-Whisker-Plots:

Visit "Early Tx DC (TXDC)" denotes Early Treatment Discontinuation Visit. Reference Ranges do not necessarily present "values of concern" in this population but will give some context to the results relative to a normal population.

#### (Notes for programmer:

- replace <Parameter> <unit>, in label by actual parameter and unit used
- Adapt Visits as relevant for the different parameters. Not all parameters are reported for all visits, only scheduled visits to be included in the Figure
- display for: Hemoglobin, Platelets, Activated partial thromboplastin time (aPTT), prothrombin time (PT), Prothrombin International Normalized Ratio (INR), d-dimer, Anti-Xa, Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Total bilirubin, Creatinine, Creatinine Clearance, Estimated)
- Include reference lines for each parameter in the Box-Whisker-Plot based on the table below. Use the last column "Proposed Reference Range for Boxplots".

Given that normal ranges for laboratory values vary from center to center, we propose standard reference lines be added to the boxplots based on ranges available from the American Board of Internal Medicine (January 2020). Specifically, we will implement this approach according to the ranges noted in the table below without objection. It should be noted that these ranges do not necessarily represent "values of concern" in this population but will give some context to the results relative to a normal population.

| Test | ABIM Reference Range | Proposed Reference<br>Range for Boxplots |
|---|---|---|
| Hemoglobin | Female: 120-160 g/L<br>Male: 140-180 g/L | 120-180 g/L |
| Platelets | 150-450 10^9/L | 150-450 10^9/L |
| aPTT | 25-35 sec | 25-35 sec |
| PT | 11-13 sec | 11-13 sec |
| PT-INR* | n/a | 0.8-1.2 |
| D-dimer | <0.5 mg/L | 0-0.5 mg/L |
| Anti-Xa | 0.3-0.7 IU/mL | 0.3-0.7 IU/mL |
| AST | 10-40 U/L | 10-40 U/L |
| ALT | 10-40 U/L | 10-40 U/L |
| Total Bilirubin | 5.13-17.10 umol/L | 5.13-17.10 umol/L |
| Creatinine | Female: 44.21-97.26 umol/L Male: 61.89-114.95 umol/L | 44.21-114.95 umol/L |
| Creatinine Clearance | 90-140 mL/min/1.73m <sup>2</sup> | 90-140 mL/min |

<sup>\*</sup> Upper reference corresponds to lowest CTCAE Grade 1 result; lower reference from Medline

Table 17: Listing of Prior and Concomitant Medications (only Targeted Medications) - Safety Set

| Subject<br>Age/Sex/Race | Treatment<br>Group | ATC Level 2/<br>Preferred Term/<br>Medication Name | Start Date<br>(Study Day) | Stop Date<br>(Study Day) | Dose<br>[Unit] | Frequency | Route | Indication |
|---|---|---|---|---|---|---|---|---|
| 999-999 /<br>70/F/W | DSTAT<br>0.25 | ATC Level 2 Preferred Term Medication Name | DdMMMyy (xx) | DdMMMyy (xx) | 40 [mg] | BID | IV | AE: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| 999-999 /<br>xx/xx/xx | Cohort 1<br>PBO | ATC Level 2<br>Preferred Term<br>Medication Name | DdMMMyy (xx) | Ongoing | | | PBO | MH: xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| 999-999 /<br>xx/xx/xx | Cohort 1<br>PBO | ATC Level 2 Preferred Term Medication Name | DdMMMyy (xx) | Ongoing | | | PBO | PR: xxxxxxxx |

Note: Medications are coded using WHO-DD Version March 2020.

Study Days prior to first treatment date are calculated as (actual date - first treatment date), after first treatment date as (actual date - first treatment date) + 1.

AE: Adverse Event, MH: Medical History, PR: Prophylaxis or Other

Page x of y

```
(Notes for programmer:
```

- Sorted by subject number, start date, stop date, ATC Level 2, preferred term and Medication Name
- Target Medications are:

Remdesvir (WHO-DC starting with "142690")
Dexamethasone (WHO-DC starting with "000160")

Anti-XA (enoxaparin) (WHO-DC starting with "017082" or "000277")

- Indication: If multiple, concatentate and wrap, drop the AE/MH-Numbers

This document is confidential.

#### 5.2. ADDITIONAL POST-COHORT 2 LOCK ANALYSES - TABLE SHELLS

Figure 4: Biomarkers during the course of the study - Safety Set

```
Line-plots
Biomarker: <HMGB1 (SI-unit)> <IL-6 (SI-unit)> <TNF alpha (SI-unit)> - see list of Biomarkers on the next page
y-axis:
       range: depending on data
       label: Value (unit)
x-axis:
       range: Baseline (D1), Day 3 (D3), Day 5 (D5), Day 7 (D7), Day 14 (D14), Day 28 (D28)
       label: Visit
       Line-Plots: different line styles/colors to differentiate cohort/group
Lines:
       one line per subject
       4 different line styles/colors to differentiate cohort/group
(Notes for programmer:
- one figure per biomarker,
- additional Biomarkers might be added on short notice of sponsor
- "(SI-unit) » in sub-title to be replaced by actual SI-unit
See list of Biomarkers provided by Chimerix on 9Dec2020
```

| 25964 | SAA,EDTApl(-70)RUO387PNL | ng/mL | ng/mL | Biomarkers |
|---|---|---|---|---|
| 25965 | IL-6,EDTApl(-70)RUO387PNL | pg/mL | pg/mL | Biomarkers |
| 25966 | TNF-alpha,EDTAp1(-70)RUO387PNL | pg/mL | pg/mL | Biomarkers |
| 26776 | AT-III,EDTApl(-80)RUO387 | ug/mL | ug/mL | Biomarkers |
| 26777 | Ficolin-3,EDTApl(-80)RUO387 | ug/mL | ug/mL | Biomarkers |
| 5592 | GM-CSF, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5593 | IFN-gamma,EDTAp1(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5594 | IL-10, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5615 | IL-18, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5597 | IL-2, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Bio markers |
| 5632 | IL-3, EDTApl(-80)RUO-387 | ng/mL | ng/mL | Biomarkers |
| 5627 | IL-4, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5598 | IL-5, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5617 | IL-7, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5600 | IL-8, EDTAp1(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 26778 | LRG1,EDTApl(-80)RUO3 87 | ug/mL | ug/mL | Bio markers |
| 5623 | MIP1 alpha, EDTAp1(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5624 | MIP-1b, EDTAp1(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 5619 | MCP-1, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 26779 | Nr-CAM,EDTApl(-80)RUO387 | ng/mL | ng/mL | Biomarkers |
| 26780 | Neuropilin-1,EDTApt(-80)RUO387 | ng/mL | ng/mL | Biomarkers |
| 26781 | NAP-2,EDTApl(-80)RUO387 | ng/mL | ng/mL | Bio markers |
| 26782 | PEDF,EDTApl(-80)RUO387 | ng/mL | ng/mL | Biomarkers |
| 26783 | RAGE,EDTApl(-80)RUO387 | ng/mL | ng/mL | Biomarkers |
| 26784 | \$HBG,EDTApl(-80)RUO387 | nmol/L | nmol/L | Biomarkers |
| 26785 | Sortilin,EDTApl(-80)RUO387 | ng/mL | ng/mL | Biomarkers |
| 26786 | \$OD-1,EDTApl(-80)RUO387 | ng/mL | ng/mL | Biomarkers |
| 26787 | TAFI,EDTApl(-80)RUO387 | ug/mL | ug/mL | Biomarkers |
| 5626 | TNF beta, EDTApl(-80)RUO-387 | pg/mL | pg/mL | Biomarkers |
| 8966 | HMGB1,K3EDTApl(-70)RUO639 | pg/mL<br>pg/mL | pg/mL | Biomarkers |

Table 18: Proportion of and time to invasive mechanical ventilation or all-cause mortality - ITT Set

| | DSTAT 0.25<br>N=xxx | Cohort 1 PBO<br>N=xxx | DSTAT 0.325<br>N=xxx | Cohort 2 PBO<br>N=xxx |
|---|---|---|---|---|
| Number of subjects who are alive and free of invasive mechanical ventilation or ECMO through Day 28 (a) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of subjects with any invasive mechanical ventilation, ECMO, all-cause mortality or early study discontinuation, whatever comes first, n (%) (b) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any invasive mechanical ventilation, ECMO | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Early study discontinuation < Day 25 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| <pre>Kaplan-Meier estimates (c) Number of censored subjects, n (%) (c)</pre> | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to first invasive mechanical ventilation, ECMO or all-cause mortality (days) (c) | | | | |
| 25% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| Median (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| 75% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; ECMO: Extracorporeal membrane oxygenation.

- (a) Early study discontinuation before Day 25 are not included.
- (b) Subjects with any invasive mechanical ventilation, ECMO, all-cause mortality or early study discontinuation before Day 25 will be counted as event.
- (c) Kaplan-Meier estimates: Subjects with any invasive mechanical ventilation, ECMO or all-cause mortality will be counted as event. All other subjects will be censored. Time to first invasive mechanical ventilation, ECMO or all-cause mortality, whatever comes first (days): Days are calculated as (start date/time first study drug date/time)/24h). Time will be censored at last individual date/time reported. If time is not available for events "00:01" will be imputed, for censored observations "23:59" will be imputed. Randomized untreated subjects will be censored at time = 0.

Page X of Y

```
(Notes for programmer: Subjects randomized not treated will be counted in
    a) as failure, and therefore not included in (a)
    b) as event (in the line "Early study discontinuation < Day 25") in case of early study discontinuation < Day 25
    c) as censored observation (censor time = 0)</pre>
```

Figure 5: Time to invasive mechanical ventilation, ECMO or all-cause mortality (KM-Plot) - ITT Set

```
Kaplan-Meier Plot:
v-axis:
       range: 0% to 100% by 20%
       label: Event-free Probability
       reference-line: 50%
x-axis:
       range: 0 to xxx (depending on data), by 7 days
       label: Time to Event (Days)
Lines:
       solid
       different colors/line styles for the treatment-groups
       starting at (100%/Baseline)
       Censored values marked
Footnote:
N = Number of subjects in a specific group; (+) = censored values;
Kaplan-Meier estimates: Subjects with any invasive mechanical ventilation, ECMO or all-cause mortality will be counted as event.
All other subjects will be censored.
Time to first invasive mechanical ventilation, ECMO or all-cause mortality, whatever comes first (days): Days are calculated as
(start date/time - first study drug date/time)/24h). Time will be censored at last individual date/time reported. If time is not
available for events "00:01" will be imputed, for censored observations "23:59" will be imputed. Randomized untreated subjects will
be censored at time = 0.
(Notes for programmer: Subjects randomized not treated will be counted as censored observation (censor time = 0)
```

Table 19: Proportion of and time to all-cause mortality - ITT Set

| | DSTAT 0.25<br>N=xxx | Cohort 1 PBO<br>N=xxx | DSTAT 0.325<br>N=xxx | Cohort 2 PBO<br>N=xxx |
|---|---|---|---|---|
| Number of subjects with all-cause mortality or early study discontinuation, n (%) (a) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Early study discontinuation < Day 25 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Kaplan-Meier estimates (b) | | | | |
| Number of censored subjects, n (%) (b) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to all-cause mortality (days) (b) | | | | |
| 25% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| Median (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| 75% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N;

Page X of Y

(Notes for programmer: Subjects randomized not treated will be counted in

a) as event (in the line "Early study discontinuation < Day 25") in case of early study discontinuation < Day 25

b) as censored observation (censor time = 0)

<sup>(</sup>a) Subjects with all-cause mortality or early study discontinuation before Day 25 will be counted as event.

<sup>(</sup>b) Kaplan-Meier estimates: Subjects who died will be counted as events. All other subjects will be censored. Time to all-cause mortality (days): Days are calculated as (start date/time - first study drug date/time)/24h). Time will be censored at last individual date/time reported. If time is not available for events "00:01" will be imputed, for censored observations "23:59" will be imputed. Randomized untreated subjects will be censored at time = 0.

Figure 6: Time to all-cause mortality (KM-Plot) - ITT Set

```
Kaplan-Meier Plot:
y-axis:
       range: 0% to 100% by 20%
       label: Event-free Probability
       reference-line: 50%
x-axis:
       range: 0 to xxx (depending on data), by 7 days
       label: Time to Event (Days)
Lines:
       solid
       different colors/line styles for the treatment-groups
       starting at (100%/Baseline)
       Censored values marked
Footnote:
N = Number of subjects in a specific group; (+) = censored values;
Kaplan-Meier estimates: Subjects who died will be counted as event. All other subjects will be censored.
Time to all-cause mortality (days): Days are calculated as (start date/time - first study drug date/time)/24h). Time will be
censored at last individual date/time reported. If time is not available for events "00:01" will be imputed, for censored
observations "23:59" will be imputed. Randomized untreated subjects will be censored at time = 0.
(Notes for programmer: Subjects randomized not treated will be counted as censored observation (censor time = 0)
```

Table 20: Proportion of participants who are alive, discharged from the hospital, and not using home oxygen - ITT Set

| Visit | DSTAT 0.25<br>N=xxx | Cohort 1 PBO<br>N=xxx | DSTAT 0.325<br>N=xxx | Cohort 2 PBO<br>N=xxx |
|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) |
| Day 8 (D8) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 14 (D14) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 28 (D28) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in a specific group; n = Number of subjects with data available;

Subjects who discontinued study early prior to start of time window (-3 days to -1 day for each visit) will be considered as failures even if alive and last records indicate no oxygen and out of hospital.

If the discontinuation is within the time window for the respective visit the last available status to be considered.

Page X of Y

(Notes for programmer:

Number of subjects who are alive, discharged from the hospital and not using home oxygen are defined based on the Ventilator/Oxygen/Medical Care Status and the Hospitalization/Activity Status eCRF pages:

All subjects who are

- not hospitalized (either with limited activities or not) AND
- do not require oxygen (no matter whether ongoing medical care is required or not)

at the specific time points will meet this endpoint.

Use the CDISC study day - for corresponding start and stop date (e.g. hospitalization stop date, or start date of not require oxygen) and assign the relevant study days to the corresponding visit (Day 8, Day 14 and Day 28).

- Determine status on particular day with respect to death, hospitalization, and oxygen use. For example, if a subject starts oxygen (e.g. Nasal Supplemental Oxygen) on Day -1 and stops on Day 10, subject is using oxygen at Visit Day 8, subject is not using oxygen at Day 14 and Day 28.
- If can't determine one, pick the **worst status** on that day. For example oxygen stops on Day 8, subject will be considered to be on oxygen for Day 8 analysis and subject is not using oxygen at Day 14 and Day 28.

  Subject discharge from the hospital on Day 8, subject will be considered to be in the hospital for Day 8 analysis and to be discharged from the hospital on Day 14 and Day 28.
- Subjects who discontinued study early **PRIOR** to start of time window (-3 days to -1 day for each visit) will be failures even if alive and last records indicate no oxygen and out of hospital. Subjects who discontinued study early but within the time window of the respective visit, e.g. on Day 7, discharged from hospital earlier and not using home oxygen will be considered with the last available status at Day 8 (= no failure), and as failure at Day 14 and Day 28. Subjects who discontinued study early on Day 10 will be considered as failure at Day 14 and Day 28.)
- Subjects randomized not treated will be counted as failure at the respective visit in case of early study discontinuation prior to start of the time window (-3 days to -1 day for each visit).

Table 21: Clinical status assessed by the NIAID ordinal scale at fixed time points - ITT Set

| Visit | DSTAT 0.25 | Cohort 1 PBO | DSTAT 0.325 | Cohort 2 PBO<br>N=xxx |
|---|---|---|---|---|
| NIAID Score | N=xxx | N=xxx | N=xxx | |
| | n (%) | n (%) | n %) | n (%) |
| Day 8 (D8) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 14 (D14) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Day 28 (D28) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Missing | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; NIAID scores are derived according to Appendix 4 of the study protocol. Higher values indicates a better outcome. For subjects who discontinued study early within the time window (-3 days to - 1 day for each visit), the last available NIAID scale will be used at the corresponding visit and a NIAID score = missing to be assigned to all visits after early study discontinuation date.

Page X of Y

(Notes for programmer:

Use a skeleton and include all 8 NIAID scores in the table for each visit and include Missing category)

The NIAID ordinal score at the predefined time points will be derived based on the eCRF data collected on the Ventilator/Oxygen/Medical Care Status, the Hospitalizations/Activities Status pages and the death date. In the event subjects transition from one score to another on a particular Day, the worse score will be used.

Use the CDISC study day - for corresponding start and stop date (e.g. hospitalization stop date, or start date of nasal suppplemental oxygen) and assign the relevant study days to the corresponding visit (Day 8, Day 14 and Day 28).

- Determine status on particular day with respect to death, hospitalization, and ventilatory care status. For example, if a subject starts nasal supplemental oxygen on Day -1 and stops on Day 10, and if the subject is still in hospital at Day 8, a NIAID score = 4 to be assigned at Day 8.
- If can't determine one, pick the worst status on that day.

  For example nasal supplemental oxygen stops on Day 8, and subject does not require oxygen but requires ongoing medical are starting on Day 8, and the subject is in hospital at Visit Day 8, a NIAID score = 4 to be assigned at Day 8.
- For subjects who discontinued study early within the time window (-3 days to 1 day for each visit), the last available NIAID score will be used at the corresponding visit and a NIAID score = missing will be assigned to all visits after early study discontinuation date.

  E.g. if a subject withdraw from study on Day 7, his or her last NIAID score will be assigned to Day 8, and NIAID scores at Day 14 and Day 28 are considered as missing. If subject withdrawal on Day 8, his or her Day 8 NIAID score will be assigned to Day 8, and NIAID scores at Day 14 and Day 28 are considered as missing.
- For subjects who died e.g. prior to or on Day 8 a NIAID score = 1 will be assigned for the visits on and after Day 8
- Subjects randomized not treated will be counted as missing at the respective visit in case of early study discontinuation prior to start of the time window (-3 days to -1 day for each visit).

Table 22: Time to clinical improvement - ITT Set

| | DSTAT 0.25<br>N=xxx | Cohort 1 PBO<br>N=xxx | DSTAT 0.325<br>N=xxx | Cohort 2 PBO<br>N=xxx |
|---|---|---|---|---|
| Number of participants with clinical improvement, n (%) (a) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Kaplan-Meier estimates (b) | | | | |
| Number of censored subjects, n (%) (b) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of subjects without improvement | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to clinical improvement (days) (b) | | | | |
| 25% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| Median (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| 75% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; Clinical improvement is defined as at least a 2-grade improvement from baseline on the NIAID ordinal score.

Page X of Y

(Notes for programmer: Subjects randomized not treated will be counted as censored observation (censor time = 0)

<sup>(</sup>a) Subjects with a clinical improvement will be counted as event.

<sup>(</sup>b) Kaplan-Meier estimates: Subjects with a clinical improvement will be counted as event. Subjects without a clinical improvement or deaths occurring prior to the positive event will be censored. Time to clinical improvement: Days are calculated as (start date/time - first study drug date/time)/24h). Time will be censored at last individual date/time reported. If time is not available for events "23:59" will be imputed, for censored observations "00:01" will be imputed. Participants who died prior to Day 28 without clinical improvement will be censored at Day 28. Randomized untreated subjects will be censored at time = 0.

Figure 7: Time to clinical improvement (KM-Plot) - ITT Set

```
Kaplan-Meier Plot:
y-axis:
       range: 0% to 100% by 20%
       label: Event Probability
       reference-line: 50%
x-axis:
       range: 0 to xxx (depending on data), by 7 days
       label: Time to Event (Days)
Lines:
       solid
       different colors/line styles for the treatment-groups
       starting at (0%/Baseline)
       Censored values marked
Footnote:
N = Number of subjects in a specific group; (+) = censored values;
Clinical improvement is defined as at least a 2-grade improvement from baseline on the NIAID ordinal score.
Kaplan-Meier estimates: Subjects with a clinical improvement will be counted as event. Subjects without a clinical improvement or
deaths occurring prior to the positive event will be censored.
Time to clinical improvement (days): Days are calculated as (start date/time - first study drug date/time)/24h). Time will be
censored at last individual date/time reported. If time is not available for events "23:59" will be imputed, for censored
observations "00:01" will be imputed. Participants who died prior to Day 28 without clinical improvement will be censored at Day
28. Randomized untreated subjects will be censored at time = 0.
(Notes for programmer: Subjects randomized not treated will be counted as censored observation (censor time = 0)
```

Table 23: Number of ventilator-free days from baseline through Day 28 - ITT Set

| | DSTAT 0.25<br>N=xxx | Cohort 1 PBO<br>N=xxx | DSTAT 0.325<br>N=xxx | Cohort 2 PBC<br>N=xxx |
|---|---|---|---|---|
| umber of ventilator-fre | ee days, n(%) | | | |
| 0 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 4 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 5 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 6 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 7 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 8 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| 28 | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| n | xxx | Xxx | xxx | XXX |
| Mean | XX.X | XX.X | XX.X | xx.x |
| SD | XX.X | XX.X | XX.X | xx.x |
| Median | XX | Xx | xx | xx |
| Q1, Q3 | XX, XX | xx, xx | xx, xx | xx, xx |
| Min, Max | XX, XX | XX, XX | xx, xx | xx, xx |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N; SD: Standard deviation; Q1, Q3: First, third quartile; Min: minimum; Max: maximum.

Ventilator-free days are only counted through the date of early study discontinuation, study completion date or Day 28, whichever comes first. For subjects who die during the course of the study, number of ventilator-free days is defined as 0.

Page X of Y

(Notes for programmer: Include only the categories of Days (0-28) in the table which are available in the data

Table 24: Time to last hospital discharge - ITT Set

| | DSTAT 0.25<br>N=xxx | Cohort 1 PBO<br>N=xxx | DSTAT 0.325<br>N=xxx | Cohort 2 PBO<br>N=xxx |
|---|---|---|---|---|
| Number of subjects discharged from hospital, n $(\$)$ (a) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Kaplan-Meier estimates (b) | | | | |
| Number of censored subjects, n (%) (b) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Number of subjects alive and still in hospital | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Death | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Time to hospital discharge (days) (b) | | | | |
| 25% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| Median (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |
| 75% Quartile (95% CI) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) | x.x (x.xx,x.xx) |

N = Number of subjects in a specific group; n = Number of subjects with data available; Percentages are based on N;

Time to hospital discharge (days): Days are calculated as (last hospital discharged date/time - first study drug date/time)/24h). Time will be censored at last individual date/time reported. If time is not available for events "23:59" will be imputed, for censored observations "00:01" will be imputed. Participants who died prior to hospital discharge will be censored at Day 28. Randomized untreated subjects will be censored with time to hospital discharge = 0.

(Notes for programmer: Subjects randomized not treated will be counted as censored observation (censor time = 0)

Page X of Y

<sup>(</sup>a) Subjects discharged from hospital will be counted as event.

<sup>(</sup>b) Kaplan-Meier estimates: Subjects discharged from hospital will be counted as event. Subjects who are still in the hospital or died in the hospital will be censored.

```
Figure 8: Time to last hospital discharge (KM-Plot) - ITT Set
```

```
Kaplan-Meier Plot:
y-axis:
       range: 0% to 100% by 20%
       label: Event Probability
       reference-line: 50%
x-axis:
       range: 0 to xxx (depending on data), by 7 days
       label: Time to Event (Days)
Lines:
       different colors/line styles for the treatment-groups
       starting at (0%/Baseline)
       Censored values marked
Footnote:
N = Number of subjects in a specific group; (+) = censored values;
Kaplan-Meier estimates: Subjects discharged from hospital will be counted as event. Subjects who are still in the hospital or died
in the hospital will be censored.
Time to hospital discharge (days): Days are calculated as (last hospital dischared date/time - first study drug date/time) /24h).
Time will be censored at last individual date/time reported. If time is not available for events "23:59" will be imputed, for
censored observations "00:01" will be imputed. Participants who died prior to hospital discharge will be censored at Day 28.
Randomized untreated subjects will be censored with time to hospital discharge = 0.
(Notes for programmer: Subjects randomized not treated will be counted as censored observation (censor time = 0)
```

Table 25: Time to first hospital discharge - ITT Set

For the layout refer to Table 24

Adapt footnote:
... Time to hospital discharge (days): Days are calculated as (first hospital discharged date/time - first study drug date/time)/24h)...

Figure 9: Time to first hospital discharge (KM-Plot) - ITT Set

For the layout refer to Figure 8

Adapt footnote:
... Time to hospital discharge (days): Days are calculated as (first hospital discharged date/time - first study drug date/time)/24h)...